CLINICAL TRIAL: NCT03026309
Title: PET-MRI F-DOPA Activity in the Mesocorticolimbic System and Depressive Symptoms in the Prediction of Treatment Compatibility
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, david groshar, david groshar, Assuta Medical Center
Other Study IDs: 0112-16-ASMC
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- depressed: un medicated diagnosed with major depression and scheduled to start SSRI treatment.
  Interventions: Other: no intervantion
- healthy: healthy volunteers.
  Interventions: Other: no intervantion

INTERVENTIONS:
Other: no intervantion — no intervention is being performed, only observational evaluations.

SUMMARY:
Main objectives: Comparing levels of F-DOPA reuptake rate as an indicator for Dopamine metabolism of un-medicated Depressed patients to healthy individuals in the Mesocorticolimbic System (VTA-NAc-PFC) and assessing structural differences between the two groups in the Hippocampus, Hypothalamic-Pituitary gland and Mesocorticolimbic System (VTA-NAc-PFC) and resting state fMRI.

Secondary objectives: 1. Comparing the differences of DNA Methylation in the plasma and serum of patients compared to healthy controls. 2.Assessing the correlation between symptoms' severity score (evaluated based on Hamilton Rating Scale) at base line and 6 months following treatmnt to PET 18F-DOPA uptake repertoire in the Mesocorticolimbic System, structural measurements and DNA Methylation.

Methodology: Study Design: A prospective, pilot study. 30 un medicated Depressed patients and 30 Healthy volunteers will perform a [18F] FDOPA PET/MRI scans following a HAM-D questionnaire (Hamilton rating scale of depression) and blood tests.

PET-MR (Biograph mMR, Siemens AG, Erlangen, Germany) scans will be performed using the tracer of dopamine precursor 3,4-dihydroxy-6-[18F]-fluoro-l-phenylalanine ([18F] FDOPA) that reflects L-dopa transport, L-aromatic amino acid decarboxylase activity, vesicular uptake and the number of dopamine nerve terminals. Measurements of dynamic F-DOPA parameters (Ki) and quantitative measurements of static F-DOPA ( SUVmax and SUVmean) will be performed in the ventral tagmental area (VTA), nucleus accombens (NAc) and pre-frontal cortex (PFC)which comprise the Mesocorticolimbic System, bilaterally. MRI sequences of T1, T2 3D measurements (assessing Volume) of the hippocampus, Hypothalamic-Pituitary gland and Mesocorticolimbic system, DTI measurements in the mesocorticolimbic dopaminergic tract and BOLD (resting-state f-MRI) in those brain networks. whole genome DNA Methylation from whole blood will be performed.

To date there is no quantative standard of care evaluation tool that serves psychiatrists when assigning medication for newly diagnosed depressed patients. The manner in which medications are assigned are threw symptom evaluation and trial and error. Only a third of the patients achieve remission after the first line of treatment. SSRI's are most common type of medication used to treat Major Depression today. One third of patients remains un responsive even after the fourth line of treatment (of different types of medications). Anti depression medications way of action requires time to reach its effect and in many patients with no avail or even causing symptom's severity. The PET-MR multimodality imaging tool offers a cutting edge technology ideally fitted to measure brain disorders. The use of F-DOPA radio-ligand with the PET-MR constitutes a novelty in the imaging of the depressed brain. Dopamine is one of three of the monoamine neurotransmitters targeted by anti-depressive medication, sharing metabolistic agents. dopamine has been proven to be connected to the processing of emotion, motivation, hedonism and reward threw its action in the Meso-cortico-limbic system. Epigenetics is a regulatory system that determines gene expression. It is heritable in the one hand and reacts to environmental changes on the other. It has been shown to be involved in psychiatric disorders.

PET-MR scans will be performed. DNA samples will be extracted from subject's whole blood samples taken prior to scans. Then it will be analyzed for whole genome DNA methylation. Taken together this novelty imaging technique and epigenetic mapping of peripheral markers can be used to better understand and personalize anti-depressive treatment compatibility.

DETAILED DESCRIPTION:
Introduction:

Major depressive disorder (MDD) is a versatile psychiatric disorder with a prevalence of 8-12 % of the population in many countries.

According to current approach MDD is characterized by lowered activity of monoamine neurotransmitters, it is undetermined whether it is as a result of differences in sensitivity of their receptors or depletion in the synaptic cleft due to low expression or mao-a/mao-b hyperactivity.

Most antidepressant medication used today are based on the monoamine depletion theory of depression. These medications include selective serotonine reuptake inhibitors (SSRIs), serotonine norepinephrine reuptake inhibitors (SNRI's) or Tricyclics anti-depressants (TCAs), all of which inhibit the reuptake of some or all of these monoamines, inducing elevated levels in the synaptic cleft. Some medications affect the monoamines receptors directly.

Dysfunctional dopamine neurotransmission has an essential role in deficits with attention, motivation and anhedonia which are core symptoms of depressive disorder. Pre-synaptic D2r (Dopamine 2 receptor) density in the pre frontal cortex (PFC) has shown to be significantly lower in depressed patients versus healthy individuals.

At present, most studies using imaging techniques in depressed patients use mainly different types of magnetic resonance imaging (MRI) or separate nuclear medicine imaging with positron emission tomography (PET) tracers. The role of traditional MRI in the evaluation of depression and other psychiatric disorders, in different studies, is aimed mainly to differentiate structural features and therefore help strengthening the diagnosis in that aspect. There are several structural changes measured in the brains of MDD patients compared to controls. Among them decreased hippocampal volume shown also compared to remitted patients, increased Hypothalamic-Pituitary gland volume, decreased Pre Frontal Cortex (PFC) and Basal-Ganglia volume. These findings are also established in accordance to the largest meta-analysis study of structural changes using MRI and CT scans performed to date. PET scans give indications regarding brain's general or agent specific metabolism. Most PET scans performed on depressed patient uses FDG or 11-C Serotonine radioligands. Only a few studies examine F-DOPA PET uptake in depressed patients, mostly with Parkinsonian depression and one with affective flattening or impulsive symptoms on a very small sample size (n=6). Most of the studies showing indication of decreased DOPA uptake in the striatum specifically in the Nucleus Accombens (NAc). Additional information is required indicating F-DOPA uptake in relevant regions of the brain in MDD. To the best of our knowledge this will be the first study using [18F] F-DOPA PET/MRI in depressed patients. PET/MRI offers true multimodality imaging by combining anatomy, function and molecular processes that will allow more accurate identification of disease assessment.

A fact that is well established is that genetic factors together with environmental factors occurring across the lifespan likely underlie the vulnerability for depression. However in a mega-analysis of several genomewide association studies (GWAS), which analyzed 1.2 million autosomal and X chromosome single-nucleotide polymorphisms (SNPs) found no SNP achieving genome-wide significance. This discrepancy between the consistently observed substantial heritability of major depression(18) and the fact no specific genetic variants have been identified to robustly contribute to the disorder suggests other mechanisms at work. Epigenetics refers to the changes in chromatin structure that underlies changes in gene expression and that are not associated with alterations in DNA sequence. DNA methylation is one of the systems underlies epigenetics. Methylation of the DNA requires the addition of a methyl group at the 5' position of cytosines in CpG dinucleotides. Following cytosine methylation, access of transcription factors to regulatory elements is reduced due to steric interference. DNA methylation patterns are hereditable on the one hand and dynamically react to the environment in the other hand. This trait of Epigenetics makes it a regulatory mechanisms, determining gene expression, that is congruent to the nature of psychiatric disorders. Diverse patterns of DNA methylation is observed in different tissues subjected to different environments. It is even different between separate brain regions. An Epigenome-wide association studies (EWAS) are on there way. In one of them in PFC tissue of post mortem depressed subjects researchers found enrichment in neuronal growth and developmental genes sites such as Brain drived neurotrophic factor .(BDNF) Decreased BDNF levels are a well established marker for depression. Lower levels of BDNF protein have also been reported in the hippocampus of animals exposed to chronic stress. Interestingly, administration of antidepressants increased hippocampal BDNF, preventing the stress-induced decrease. These findings are intriguing given the hippocampal volume loss observed in mood disorders and decreased BDNF serum levels in individuals with mood disorders or depressive personality traits. Based on these convergent preclinical and clinical data, the BDNF gene represents a logical target for genetic investigations of mood disorders.

Another Epigenome-wide association study analyzing whole blood DNA found IL-6 and C-reactive protein (CRP) plasma levels were increased in those persons with lifetime depression, and among those with depression only, IL-6 methylation showed an inverse correlation with plasma IL-6 and CRP.

To date there is no common imaging practice in the psychiatric clinic allowing differentiating which medicated therapy is optimal for which patient. To the best of our knowledge, this will be the first study to evaluate treatment compatibility using the combination of [18F] F-DOPA PET/MRI imaging and symptoms assessment pre-treatment.

Study Objectives and Purpose:

The aim of the study is to assess the feasibility of the modality imaging and symptom evaluation in the prediction of treatment compatibility. Dopamine metabolism measured in the mesocorticolimbic system (VTA-NAc-PFC) by 18F-FDOPA PET with structural and functional MR findings in patients diagnosed with depression pre-treatment.

Main objectives:

1. Comparing naïve levels of F-DOPA reuptake in healthy individuals to untreated Depressed patients in the Mesocorticolimbic System (VTA-NAc-PFC) and assessing structural differences between the two groups in the Hippocampus, Hypothalamic-Pituitary gland and Mesocorticolimbic System (VTA-NAc-PFC) and resting state fMRI.

Secondary objectives:

1. Comparing the differences of DNA Methylation in the plasma of patients compared to healthy controls.
2. Assessing the correlation between symptoms' severity score (evaluated based on Hamilton Rating Scale) at base line and after 6 months to PET 18F-DOPA uptake repertoire in the Mesocorticolimbic System, structural measurements and DNA Methylation.

Materials and Methods:

Study Design: A prospective, pilot study.

Clinical assessment:

A quantitative measure of symptoms' burden will be determined threw clinical assessment based on "Hamilton Rating Scale for Depression" and based on DSM-V criteria at baseline (pre-treatment), 3 months and 6 months after treatment initiation. According to DSM-5 the diagnosis of depression requires five (or more) of the following symptoms that are present during the same 2-week period and represent a change from previous functioning: (1) depressed mood (2) loss of interest or pleasure. (3) Significant weight loss or weight. (4) Insomnia or hypersomnia . (5) Psychomotor agitation or retardation.(6) Fatigue or loss of energy nearly. (7) Feelings of worthlessness or excessive or inappropriate guilt.(8) Diminished ability to think or concentrate. (9) Recurrent thoughts of death.

Symptom evaluation of Hamilton Rating Scale will be done by a psychiatrist. Finally we will attempt to link specific clusters of symptoms to treatment compatibility in accordance to imaging and molecular findings. The compatibility of treatment with these medication will be compared to percentage of treatment success in the clinic in a 'standart of care' manner. Assessment of the patient's progress will be determined by change in symptoms and/or a second scan through follow up visits after 3,6 month.

.Imaging diagnostic PET/MR protocol: We would use the evaluation of the dopamine precursor 3,4-dihydroxy-6-[18F]-fluoro-l-phenylalanine ([18F] FDOPA) uptake rate constant (K(i)) that reflects L-dopa transport. L-aromatic amino acid decarboxylase activity, vesicular uptake and the number of dopamine nerve terminals. we would like to measure and compare the [18F] F-DOPA uptake in the Mesocorticolimbic network in depressive unmedicated patients and healthy individuals. We will then examine [18F] F-DOPA uptake repertoire and characterize a typical spatiotemporal pattern along different depressive brains in accordance to the many kinds of symptoms' manifestation and molecular and demographic data. In addition, we would implement, new MR sequences such as diffuse tensor imaging (DTI) and susceptibility-weighted imaging (SWI) to evaluate the mesocoticolimbic dopaminergic tract and use T1, T2 sequences to measure Hippocampal and Hypothalamic-Pituitary gland volumes in these patients compared to healthy individuals. Furthermore we will use T2* sequence to evaluate resting state Blood-Oxygen-Level Dependent (BOLD) contrast imaging. In addition scan results will be correlated to clinical evaluation of symptoms unmedicated patients.

All scans will be performed in the department of Nuclear Medicine at Tel-Aviv Assuta Medical Center using a PET/MR scanner (Biograph mMR, Siemens AG, Erlangen, Germany) in accordance with the manufacturer's guidelines.

Patients are required to fast at least 4 hours prior to arrival to the department. Upon arrival an intravenous catheter will be placed for radiopharmaceutical and gadolinium administration. Patients will receive an intravenous injection of 10 mCi of 18F-FDOPA on the PET MR table and scanning will begin immediately. Dynamic PET parameters will be acquired along with the different MR sequences. MR of the brain will include the following sequences: T1, T2 and T2 fluid attenuated inversion recovery sequence (FLAIR), susceptibility-weighted sequences (SWI), Diffuse Tensor Imaging (DTI), blood-oxygenation level-dependent (BOLD) signals for resting-state functional imaging. In addition, perfusion of the brain will be evaluated with and without gadolinium. Aa anatomical stereotactic map of the brain will be layered in congruence to the scans using ExploreDTI Software.

For contrast-enhanced sequences we use Dotarem (gadoteric acid) (0.2 ml/kg ,0.1 mmol/kg at 2ml/s, 20ml saline flush) The total scan time will be about 45 minutes.

Data collection and procedures:

For eligible healthy volunteers, the following data will be recorded at baseline:

1. Baseline parameters: date of birth, sex, socioeconomic status, ethnicity, smoking, alcohol consumption.
2. Detailed medical history.
3. List of medications
4. Symptom's Evaluation using Hamilton Rating Scale for Depression
5. Blood sample

For eligible depressed patients, the following data will be recorded at baseline, after 3 months and after 6 months.

1. Baseline parameters: date of birth, sex,
2. Detailed medical history.
3. List of medications
4. Symptom's Evaluation using Hamilton Rating Scale for Depression
5. Blood sample
6. Clinical diagnosis and symptoms onset.

Biological Sample collection:

Blood samples will be drawn from patients and healthy controls prior to scans for the assessment of Whole genome DNA methylaion in plasma of peripheral blood. Blood samples will be taken on from healthy controls and depreesed patients on base line. From depressed subjects ,blood will be drawn olso after 6 months of treatment start date for the evaluation of gene expression mRNA or protein of specific markers based on epigenetic findings from base line.

Analysis of genome-wide promoter DNA methylation:

The procedure used for MeDIP analysis was adapted from previously published protocols.(13,14) Brieﬂy, 2μg of DNA is sonicated, and methylated DNA is immunoprecipitated using anti-5-methyl-cytosine (Eurogentec, Fremont, CA, USA). The DNA-antibody complex was immunoprecipitated with protein G, and the methylated DNA is then resuspended in digestion buffer (50mM TRisHCl pH8; 10mM EDTA; 0.5% SDS) and treated with proteinase K overnight at 55°C. The input and bound fraction is puriﬁed, ampliﬁed using the Whole Genome Ampliﬁcation Kit (Sigma-Aldrich, St. Louis, MO, USA), and labeled for microarray hybridization with Cy3-dUTP and Cy5-dUTP, respectively, using the CGH Enzymatic Labeling Kit (Agilent Technologies, Mississauga, ON, Canada) in accordance with the manufacturer´s instructions. Custom designed tiling arrays were used (Agilent Technologies). All steps of the hybridization, washing, scanning and feature extraction procedures is performed in accordance with the Agilent Technologies protocol for chipon-chip analysis. Extracted microarray intensities is processed and analyzed using the R software environment for statistical computing (http://www.r-project.org/).

Gene-speciﬁc Validation:

validation of MeDIP data will be performed applying quantitative-real time PCR (QPCR) using the 2-ΔΔCt method. Data will be expressed as group means±s.e.m. The Graphpad 5 software will be used to perform one-tailed Mann-Whitney U-tests.

RNA extraction from human blood:

blood for RNA extraction will be collected before injection of the radioligand and drawn into PAXgene Blood RNA tubes (PreAnalytiX, Hombrechtikon, Switzerland). RNA is extracted using the PAXgene Blood RNA Kit (Qiagen). The quality and quantity of RNA samples will be analyzed using an Agilent 2100 Bioanalyzer (Agilent Technologies, Böblingen, Germany).

Analysis of gene expression in human blood:

Reverse transcription will be performed using the high-capacity cDNA Reverse Transcription Kit (Life Technologies, Darmstadt, Germany). Gene expression levels will be analyzed using QPCR and the 2-ΔΔCt method. Data will be expressed as group means±s.e.m. Statistical signiﬁcance will be tested using one-tailed Mann-Whitney U-tests.

Pyrosequencing:

The promoter region of specific genes will be analyzed by pyrosequencing. In brief, fragments of bisulﬁte-treated DNA(EpiTect Bisulﬁte Kit, Qiagen) will be ampliﬁed by PCR (HotStar Taq DNA Polymerase, Qiagen) primer information using an unmodiﬁed forward primer and a biotin-labeled reverse primer (Euroﬁns, Ebersberg, Germany). Pyrosequencing will be performed using a PyroMark Q24 Advanced system (Qiagen; primer information see Supplementary Table S2) in accordance with the manufacturer's protocol. Methylated and unmethylated EpiTect control DNA samples (Qiagen) will be used as controls for bisulﬁte conversion, ampliﬁcation and pyrosequencing. The percentage of methylation at each CpG site will be quantiﬁed using the PyroMark Q24 Advanced software version 3.0.0 (Qiagen) Sequencing will be performed in triplicate. Quality control ﬁltering and statistical analyses of the pyrosequencing results will be conducted using R Version 2.15.3 (http://www.r-project.org). Measurements marked as unreliable by the Pyromark software will be removed from the data set. Triplicate measurements will be averaged after the removal of outliers (values deviating more than 3%). A Mann-Whitney U-test will be used to compare the mean percentage of methylation of CpG sites for the ELS versus control groups. Data will be presented as the mean±s. e.m.

Genetic analysis:

Genotypes will be investigated using GWAS data of a previous study of MDD. dbSNP of chosen genes (http://www.ncbi.nlm.nih.gov/projects/SNP) will be searched for SNPs (single-nucleotide polymorphisms) across the genes. The setbased test, as implemented in PLINK (v1.0.7)39 will be performed (with default options and 105 permutations), to test for association between MDD and the whole set of genetic variants in the data set

MR findings:

* T1,T2 3D measurements (assessing Volume) of the hippocampus, Hypothalamic-Pituitary gland and Mesocorticolimbic.
* DTI measurements in the mesocorticolimbic dopaminergic tract.
* Comparison of resting-state f-MRI (BOLD) brain networks in patients with depression with normal maps

PET findings:

1. Visual assessment and quantitative measurements of static F-DOPA (e.g., SUVmax and SUVmean) will be performed in the VTA, NAc, PFC bilaterally.
2. Measurements of dynamic F-DOPA parameters such as Ki when available (e.g., time to peak, peak value etc.) will be measured.

Statistics:

Patient characteristics will be summarized using descriptive statistics. Quantitative variables will be presented as mean and SD, qualitative variables will be presented as frequencies.

Pearson correlation coefficient will be used to measure the strength of the relationship between the PET in the different brain areas and the cluster symptoms.

A t-test will be used to compare the mean values of the different parameters. Sample size: This is a pilot study for which a sample size of 60 subjects (30 healthy individuals and 30 patients) is required.

Participant Sampling: All patients fulfilling inclusion criteria and providing informed consent will be consecutively enrolled.

Confidentiality:

All the data will be coded and subject will be identified only by the subject's initials and by the subject's study number.

The coding will be done by the investigators and will be saved on their secured computers and in the investigator file locked in a closet in the principal investigator office.

All reports and communications relating to subjects in the study will be using the code given, with no personal information.

ELIGIBILITY:
* Control group-30 healthy individuals:

Inclision criteria:

1. Adult male patients between the age of 30-50 years old.
2. Willing to participate and able to give there informed consent

Exclusion Criteria:

1. women.
2. With no history of psychiatric diagnosis.
3. History of any neurodegenerative disease or active oncologic disease.
4. With no history of psychiatric medication intake.
5. Patients treated with levodopa or any other medication known to interfere with the DAT or catechol O-methyltransferase inhibitors, or with dopamine receptor blocking / or catecholamine re-uptake blocking properties.
6. Contraindication to MR imaging.

study group- 30 Newly diagnosed depressed patient from the clinic of Dr. Lurie an extension of Shalvata Mental health center .

Inclusion criteria:

1. Adult male patients between the age of 30-50 years old.
2. Patients willing to participate with all the study procedures and sign informed consent form.
3. A clinical diagnosis of major depression.
4. With no history of psychiatric medication intake.
5. Scheduled to be treated with SSRI.

Exclusion criteria:

1. women.
2. Psychiatric patients diagnosed and treated with any psychiatric medication.
3. History of any neurodegenerative disease or active oncologic disease.
4. Patients with history of other brain disorder/pathology.
5. Patients treated with levodopa or any other medication known to interfere with the DAT or catechol O-methyltransferase inhibitors, or with dopamine receptor blocking / or catecholamine re-uptake blocking properties.
6. Contraindication to MR imaging.
7. With suicidal symptoms.

Subject withdrawal criteria:

1. Subject who withdrawn his consent at any point of the study.
2. Inability to perform MR
3. Non compliant with treatment intake or follow up observations.
4. Any decision made by the investigator that termination is in subject's best intrest.
5. Serius adverse event relating to the study.

   -

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sample size: This is a pilot study for which a sample size of 60 subjects (30 healthy individuals and 30 patients) is required.
  Participant recruitment:
  Eligible consecutive patients, satisfying the inclusion/exclusion criteria, will be identified and recruited by the psychiatric clinic.
  Eligible healthy volunteers will be recruited with assigned pamphlet approved by IRB.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
3,4-dihydroxy-6-[18F]-fluoro-l-phenylalanine ([18F] FDOPA) uptake rate constant (K(i)) that reflects L-dopa transport. | at base line

IPD SHARING:
Plan to Share IPD: No